CLINICAL TRIAL: NCT04931355
Title: A Randomized Controlled Study on the Short-term Intervention of Acupuncture in the Freeze-all IVF Cycle to Improve Pregnancy Rate
Brief Title: Acupuncture in the Freeze-all IVF Cycle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00006761-M2020443
Record Dates: First submitted 2021-06-15; First posted 2021-06-18 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-01

CONDITIONS: Acupuncture; Female Infertility
Keywords: Acupuncture; Traditional chinese medicine; freeze-all IVF cycle; Embryo Transfer
MeSH Terms: conditions — Infertility, Female | interventions — Acupuncture Therapy; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture treatment group (Experimental): Method: Acupuncture at Zhongwan、Qihai、Guanyuan、Zhongji、Guilai、Shenshu、Ciliao、Xuehai、Sanyinjiao、Taixi. The acupuncture treatment starts on the 5th day of the menstrual cycle and lasts to the days before IVF-ET
  Interventions: Other: Acupuncture
- Western medicine group (Active Comparator): The western medicine group will be treated with conventional western medicine
  Interventions: Other: Western medicine

INTERVENTIONS:
Other: Acupuncture — The Acupuncture intervention（Zhongwan、Qihai、Guanyuan、Zhongji、Guilai、Shenshu、Ciliao、Xuehai、Sanyinjiao、Taixi.） will start on the 5th day of menstruation cycle, which will be carried out 1 time per day, at least 5 times a week, lasts for 10-15days. All operations were performed by experienced acupuncturists. After ET, both the control group and the treatment group will be treated with conventionally with no TCM intervention.
  Other Names: conventional western medicine(Recombinant Human Follitropin Alfa for Injection、Fructose Injection、Tetyacycline Hydrochloride Capsules、Cetrorelix Acetate Powder for Injection )
  Arms: Acupuncture treatment group
Other: Western medicine — Western medicine
  Arms: Western medicine group

SUMMARY:
In the early stage, our team found that Acupuncture intervention in freeze-all IVF cycles can improve the clinical pregnancy rate. In order to further study the role of Acupuncture in improving the pregnancy outcome of IVF-ET in infertility. A randomized controlled clinical trial will be used in this study. 90 infertile patients are randomly divided into two groups. The control group will be treated with conventional modern medicine, and the treatment group will be treated with Acupuncture on the basis of conventional modern medicine. The intervention starts from the 5th day of the menstrual cycle and lasts to the day before IVF-ET. The number of oocytes, antral follicles, AMH, serum FSH, and clinical pregnancy rate will be observed to evaluate the effect of Acupuncture on the improvement of pregnancy outcome. In addition, all of the participants will be asked to complete the self-evaluation of the anxiety/depression scale on the 7th day of the menstrual cycle, before and after transplantation, to analyze the emotional changes of the subjects during the study. We observe the safety and health economic indicators of Acupuncture treatment, so as to improve the overall efficacy of TCM Combined Application in assisted reproductive technology in the future.

DETAILED DESCRIPTION:
The study will be conducted on patients with DOR attending our reproductive medicine center for proposed IVF-ET between June 2021and December 2022.

The trial is designed as a randomized, controlled clinical trial with two groups established by 1:1 equal allocation, a treatment group with interventions using acupuncture to tonify the kidneys and regulate blood and a control group treated using conventional Western medicine.

Random numbers will be prepared by an independent third-party statistician who prepared a list of random group codes for this study. Enrolled subjects will be given a subject number during the screening process and, upon formal enrolment, will be randomly assigned to either the test or control group with a corresponding random number.

The acupoints used will be:

Zhongwan (RN12) ：The needle should be punctured for 1-1.2 inches and retained for 30 minutes.

Qihai(RN6): The needle should be punctured for 1-1.2 inches and retained for 30 minutes.

Guanyuan(RN4): The needle should be punctured for 0.8-1.2 inches and retained for 30 minutes.

Zhongji(RN3): The needle should be punctured for 0.8-1.0 inches and retained for 30 minutes.

Guilai(ST29): The needle should be punctured for 0.8-1.0 inches and retained for 30 minutes.

Shenshu(BL23): The needle should be punctured for 0.8-1.0 inches and retained for 30 minutes.

Ciliao(BL28): The needle should be punctured for 1-1.2 inches and retained for 30 minutes.

Xuehai(SP10): The needle should be punctured for 1-1.5 inches and retained for 30 minutes.

Zusanli(ST36): The needle should be punctured for 1-1.5 inches and retained for 30 minutes.

Diji(SP8): The needle should be punctured for 1-1.2 inches and retained for 30 minutes.

Sanyinjiao(SP6): The needle should be punctured for 1-1.2 inches and retained for 30 minutes.

Taixi(KI6): The needle should be punctured for 0.8-1.2 inches and retained for 30 minutes.

Baihui(DU20): The needle should be punctured for 0.5-1.0 inches and retained for 30 minutes.

Yintang(EX-HN3): The needle should be punctured for 0.5-1.0 inches and retained for 30 minutes.

The Acupuncture intervention will start on the 5th day of the menstruation cycle, which will be carried out 1 time per day,at least 5 times a week, lasts for 10-15days. All operations were performed by experienced acupuncturists. After ET, both the control group and the treatment group will be treated with conventionally with no TCM intervention.

Serum human chorionic gonadotropin (hCG) will be measured, and an hCG>30 IU will be considered to indicate biochemical pregnancy. Ultrasound monitoring will be performed 30 days after ET to calculate the clinical pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for infertility.
2. Meet the criteria for identifying kidney deficiency in TCM.
3. Patients who Planning to undergo IVF-ET for pregnancy in our center, Age ≤40 years and ≥25 years.
4. Previous embryo transfer failure ≥ 2 times.
5. Menstrual cycle is basically normal, and normal ovulation has been monitored in the past.
6. There were more than 1 blastocyst /more than 2 high-quality embryos with more than 6 cells on day 3/more than 2 high-quality embryos with more than 4 cells on day 2.
7. Consent to participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Patients with endometritis, acute pelvic inflammatory disease, mycotic vaginitis, bacterial vaginitis, adnexitis or other systemic infections.
2. It has been confirmed that there are obvious and serious other organic lesions in the reproductive organs.
3. Patients with allergic constitution
4. Infertility caused by genetic factors
5. Patients with serious primary diseases such as cardio cerebrovascular, kidney, liver and hematopoietic system and psychosis
6. A person who is unable to cooperate (such as a combination of neurological or mental illness, or a reluctance to cooperate)
7. The endometrial thickness on the day of hCG was less than 6 mm or the endometrial morphology on the day of hCG was type C
8. Those who did not agree to participate in the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate (%) | up to 6 weeks from enrollment
  Follow up by telephone calls 14days after the IVF-ET

SECONDARY OUTCOMES:
Concentration of β-human Choriogonadotropin(β-HCG) | up to 6 weeks from enrollment
  Obtained by blood sampling 14 days after the proposed IVF-ET

OTHER OUTCOMES:
Changes from Baseline concentration of Self rating Anxiety Scale (SAS) | The 5th day of menstruation、 Baseline the proposed IVF-ET、14 days after the IVF-ET
  They were completed on the 5th day of menstruation, before transplantation and the 14th day after transplantation.The score of 20 items is added to get the rough score (x), and after the formula is converted, that is, the whole part is taken after multiplying the rough score by 1.25, and then the standard score (y) will be obtained.According to the results of Chinese norm, the cut-off value of SAS standard deviation was 50 points, of which 50-59 points were mild anxiety, 60-69 points were moderate anxiety, and more than 69 points were severe anxiety.
Changes from Baseline concentration of Self rating Depression Scale (SDS) | The 5th day of menstruation、 Baseline the proposed IVF-ET、14 days after the IVF-ET
  They were completed on the 5th day of menstruation, before transplantation and the 14th day after transplantation.The normal upper limit of SDS gross score is 41, and the lower the score, the better the state. The standard is divided into the integral part of the total rough score multiplied by 1.25. In China, SDS score ≥ 50 is regarded as depressive symptom.Severity of depression = cumulative score of each item / 80. Results: no depression was found in patients below 0.5; 5-0. 59 for mild to mild depression; 6-0. 69, moderate to severe; More than 0.7 was severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China, China